CLINICAL TRIAL: NCT01426516
Title: A Six-month Study of the Genecept Assay vs. Treatment as Usual to Evaluate Efficacy of Using Assay Guided Treatment in Outpatient Adults With Treatment Resistant Depression
Brief Title: Pharmacogenomics for Antidepressant Guidance and Education 1 (PAGE-1_AG1)
Acronym: PAGE-1_AG1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Invalid data collection
Sponsor: Genomind, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AG1-0001/2
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-08

CONDITIONS: Major Depressive Disorder
Keywords: Treatment Resistant; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Genetic Testing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as usual (TAU) (No Intervention): Subjects will give DNA sample for genetic testing but will not receive genetic results and will therefore receive treatment as usual.
- Genecept Assay (Experimental): Subjects donate DNA sample for genetic testing and treatment decisions take genetic results into account.
  Interventions: Device: Genecept Assay

INTERVENTIONS:
Device: Genecept Assay — Genetic test which analyzes five pharmacodynamic and two pharmacokinetic genes important in psychiatric disorders
  Other Names: Genetic Test
  Arms: Genecept Assay

SUMMARY:
One-third or more of individuals treated for major depressive disorder (MDD) do not experience remission of symptoms despite at least two adequate antidepressant trials. Such treatment-resistant depression (TRD) contributes disproportionately to the tremendous costs of MDD, in terms of health care costs, functional impairment, and diminished quality of life.

The promise of personalized medicine for individuals at high risk for TRD is apparent. If these individuals could be recognized early in their disease course, they could be triaged to more intensive or targeted interventions to improve their likelihood of remission. With the proliferation of treatment options in MDD, at present individuals can spend months or years in and out of treatment before receiving these next-step treatments.

At present, no clinical or biomarker-based tool has been shown to assist in matching patients with treatments most likely to be effective for them. The Genecept Assay offers the possibility of "Personalized Medicine" in psychiatry. Clinicians may find this additional genetic information can lead to optimized treatment plans for individual patients. Before such an assay can be widely applied clinically, it is necessary to demonstrate that this tool usefully impacts treatment outcomes.

This study will examine the potential impact of the assay in terms of depression severity at 3 months, with further follow-up out to 6 months. Secondary measures will allow an estimate of its potential to change clinician behavior and improve patient quality of life. Further measures will also allow for refinement of the assay to maximize patient and clinician satisfaction, and estimate the potential savings associated with deployment of this assay in real-world clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* written informed consent
* diagnosis of non-psychotic major depression as determined by study
* clinician/current medical prescriber, and mood disorder diagnosis confirmed by PHQ-9
* QIDS-SR score of at least 10 (i.e., moderate depression) at initial visit
* failure of at least 1 prior adequate trial of a standard antidepressant (by ATRQ criteria - i.e., 6 weeks at adequate dose)

Exclusion Criteria:

* psychotic features in the current episode, based upon clinical assessment
* 4 or more failed pharmacologic interventions in the current major depressive episode [response rates for these subjects is likely to be extremely low and would require a substantially larger-scale study to identify treatment effects]
* current substance use disorder other than nicotine which based upon clinical assessment requires inpatient or outpatient detoxification
* pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (to include oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or partner with vasectomy)
* women who are breastfeeding
* serious suicide or homicide risk, as assessed by evaluating clinician
* other unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease, based on review of medical history, physical examination, and screening laboratory tests
* patients who have taken an investigational psychotropic drug within the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Dicker, PharmD, Study Director — Genomind, LLC
Locations (1):
- Centerstone, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment as Usual (TAU) | Genecept Assay
Started | 12 | 17
Completed | 12 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual (TAU) | Genecept Assay | Total
Number analyzed (Participants) | 12 | 17 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 17 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 44 [24 to 59] | 46 [23 to 65] | 45 [23 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 1 | 6 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 17 | 28
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Measured by Change in Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR), Adjusted for Baseline Severity, at 6 Months
Description: To determine the efficacy of assay-guided treatment (AGT) versus treatment-as-usual (TAU), in terms of depression severity as measured by change in Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR), adjusted for baseline severity, at 6 months
  Add:
  * highest score on any 1 of the 4 sleep items (items 1 to 4)
  * highest score on any 1 of the 4 weight items (items 6 to 9)
  * highest score on either of the 2 psychomotor items (15 and 16)
  * scores for each of the 6 MDD symptom domains
  Total scores range from 0-27. 0 = no signs of depression; 27 = severe depression
Time Frame: 6 months
Population: Invalid Data Collection
Arm/Group | Treatment as Usual (TAU) | Genecept Assay
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Clinician Behavior as Measured by Change in Recorded Treatment Choice Before and After the Assay Results Are Made Available.
Description: Clinicians will rank first and alternative treatment choice and dosage prior to assay and first and two alternative treatment choices after receiving assay results (for AGT group). Clinician choices will be compared.
Time Frame: one week
Population: Invalid data collection
Arm/Group | Treatment as Usual (TAU) | Genecept Assay
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quality of Life as Measured by Self Reported Assessment of Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ)
Description: To determine the efficacy of assay-guided treatment (AGT) versus treatment-as-usual (TAU) in outpatient treatment of nonpsychotic major depressive disorder, in terms of patient quality of life (Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ)) The minimum raw score on the QLESQ is 14, and the maximum score is 70.
Time Frame: baseline, 3, 6 months
Population: Invalid data collection
Arm/Group | Treatment as Usual (TAU) | Genecept Assay
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Cost
Description: To compare costs of AGT versus TAU in outpatient treatment of nonpsychotic major depressive disorder as measured by claims data.
Time Frame: 6 months
Population: invalid data collection
Arm/Group | Treatment as Usual (TAU) | Genecept Assay
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Acceptability of the Use of AGT for Subjects and Clinicians as Measured by Satisfaction Survey
Description: To determine the acceptability to patients and clinicians of assay-guided treatment (AGT) versus treatment-as-usual (TAU) in outpatient treatment of nonpsychotic major depressive disorder
Time Frame: 6 months
Population: invalid data collection
Arm/Group | Treatment as Usual (TAU) | Genecept Assay
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Treatment as Usual (TAU) | Genecept Assay
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/17
Other Adverse Events (participants affected / at risk) | 3/12 | 6/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment as Usual (TAU) (N=12) | Genecept Assay (N=17)
Minor to Moderate Adverse Effects to Medications (Psychiatric disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes